CLINICAL TRIAL: NCT07125261
Title: BHV-7000 Efficacy Against Epileptiform Activity in Patients With Epilepsy Implanted With RNS
Brief Title: BHV-7000 Responsive Neurostimulation System (RNS) Study
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Biohaven Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Imran Quraishi, Associate Professor of Neurology, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000039852
Record Dates: First submitted 2025-08-08; First posted 2025-08-15 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Epilepsy; Seizures
Keywords: neurostimulation; antiseizure medication; RNS
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Intervention Model Description: The study population includes adults with focal epilepsy who have been implanted with RNS and continue to have epileptiform activity in their RNS device recordings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BHV-7000 (Experimental): Participants will receive up to 28 days of study drug and will be followed clinically until Day 56, making their total involvement in the study up to 84 days. The study follows an ABA treatment paradigm with (A) 90-day retrospective RNS baseline, (B) 4-week treatment period, and (A) 4-week withdrawal period.
  Interventions: Drug: BHV-700

INTERVENTIONS:
Drug: BHV-700 — 75 mg daily for the 4-week treatment period (dose which may be adjusted based on tolerability)

SUMMARY:
This is an open label study to assess the biological effect of BHV-7000 on abnormal activity recorded by the RNS System in patients with focal epilepsy implanted with the RNS System. BHV-7000 is a potassium channel activator being evaluated for use in epilepsy. Participants are offered the drug for 4 weeks. Activity during that treatment period is compared to a 90-day retrospective baseline period in which other medications and device settings were stable, and also to a 4-week withdrawal period after treatment is discontinued. The study is open to patients with RNS regardless of whether they report clinical seizures, as long as the device recordings continue to show epileptiform activity.

DETAILED DESCRIPTION:
This is an open-label proof-of-principle study to assess the biological effect BHV-7000 on epileptiform activity detected by the RNS System. The study uses a single case experimental design in a small number of participants. Following a 90-day retrospective baseline period, there is a 4-week treatment period followed by a 4-week withdrawal period. Objective electrophysiologic biomarkers will be obtained from patients' RNS and analyzed in each participant to assess patient-level efficacy.

The primary objective of this study is to determine whether BHV-7000, a potassium channel activator, reduces the frequency of electrographic biomarkers of epileptic activity detected in patients with epilepsy who were implanted with the RNS System.

Secondary objectives are assess whether BHV-7000 withdrawal in participants leads to subsequent worsening of electrographic biomarkers of seizures compared to the treatment period, and to assess the safety and tolerability of BHV-7000 in participants with epilepsy who have been implanted with RNS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of focal epilepsy as documented in the medical record.
* Implanted at least 1 year ago with RNS.
* RNS device actively recording intracranial EEG data.
* Baseline RNS recordings show that the over 50% of detections represent epileptiform seizure onset patterns.
* Provision of signed and dated informed consent form.
* Ability to take oral medication and be willing to adhere to the BHV-7000 treatment regimen.
* Body mass index (BMI) < 40 kg/m² at screening visit.

Exclusion Criteria:

* Change in any antiseizure medication (including addition or discontinuation of any antiseizure
* Any change in RNS detection settings within 90 days prior to planned treatment Day 1.
* Change in RNS stimulation settings within 90 days prior to planned drug administration (retrospective baseline period).
* Poor or inconsistent history of device downloads in the 90 days prior to planned treatment Day 1, as determined by less than 90% of episode start data being available at treatment Day 1.
* RNS battery low (estimated to last for less than 3 months).
* Schizophrenia and other psychotic disorders (e.g., schizophreniform disorder, schizoaffective disorder, psychosis not otherwise specified [NOS]), bipolar disorder, and/or obsessive-compulsive disorder, or other serious mental health disorders. Uncontrolled unipolar major depression where changes in pharmacotherapy are needed or anticipated during the study.
* Active suicidal plan/intent in the past six months, a suicide attempt in the last two years, or more than one lifetime suicide attempt.
* History of illicit drug or alcohol abuse within one year prior to screening judged by the PI to be excessive or compulsive, or currently using drugs of abuse or any prescribed or over the counter medication in a manner that the PI considers indicative of abuse or dependence.
* History of cancer within the past two years, with the exception of appropriately treated basal cell or squamous cell carcinoma.
* History of clinically significant urinary retention in the judgment of the PI.
* Previous exposure to BHV-7000 or known allergy to BHV-7000 or its excipients.
* Any major surgery within one month or an acute illness within two weeks prior to screening.
* Vaccination within the previous four weeks prior to screening or planned vaccination during the study.
* History of ezogabine use.
* Known allergic reactions to components of the study drug.
* Febrile illness within 90 days prior to planned treatment Day 1.
* Significant cardiovascular history, including but not limited to uncontrolled angina, myocardial infarction (Ml) within 12 months of screening, clinically significant arrhythmia, congestive heart failure (New York Heart Association [NYHA] Class Ill or higher).
* QTcF (Fridericia) interval 450 msec for males and 470 msec for females; Mobitz Type II second or third degree atrioventricular (AV) block, or complete left bundle branch block, or complete right bundle branch block, or intraventricular conduction defect with a QRS duration 130 msec, or evidence of acute or sub-acute myocardial infarction (Ml) or ischemia, or other ECG findings that, in the investigator's opinion, would preclude participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Reduction in patient-specific seizure surrogate rate | 28 days
  Per-participant percentage reduction in patient-specific seizure surrogate rate in the treatment period relative to retrospective baseline.
Reduction in seizure onset pattern rate | 28 days
  Per-participant percentage reduction in seizure onset pattern rate in the treatment period relative to retrospective baseline.
Reduction in long episode rate | 28 days
  Per-participant reduction in long episode rate during the treatment period relative to the retrospective baseline.
Reduction in saturation rate | 28 days
  Per-participant reduction in saturation rate during the treatment period relative to the retrospective baseline, for those patients who have saturations.

SECONDARY OUTCOMES:
Withdrawal effect on patient-specific seizure surrogate rate | 4 weeks post 28-day treatment
  Change in patient-specific seizure surrogate rate following drug withdrawal.
Withdrawal effect on seizure onset pattern rate | 4 weeks post 28-day treatment
  Change in seizure onset pattern rate following drug withdrawal.
Withdrawal effect on long episode rate | 4 weeks post 28-day treatment
  Change in long episode rate following drug withdrawal.
Number of Participants With Treatment-Related Laboratory Abnormalities or Adverse Events of Special Interest (AESI) as Assessed by CTCAE/DAIDS | up to 12 weeks
  Treatment-emergent laboratory abnormalities and AESIs will be reported. Higher score corresponding to increasing AE severity.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Quraishi, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Yale Comprehensive Epilepsy Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No